CLINICAL TRIAL: NCT04842604
Title: A MULTI-CENTER CONTINUATION STUDY EVALUATING AZACITIDINE WITH OR WITHOUT GLASDEGIB (PF-04449913) IN PATIENTS WITH PREVIOUSLY UNTREATED ACUTE MYELOID LEUKEMIA, MYELODYSPLASTIC SYNDROME OR CHRONIC MYELOMONOCYTIC LEUKEMIA
Brief Title: Continuation Study of B1371019(NCT03416179) and B1371012(NCT02367456) Evaluating Azacitidine With Or Without Glasdegib In Patients With Previously Untreated AML, MDS or CMML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1371019 Open Label Extension; 2017-002822-19 (EudraCT Number)
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome; Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — glasdegib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants from B1371019 and B1371012 (Experimental): Azacitidine will be administered 75 mg/m2/day for 7 days every 28 days on Days 1-7 (±3 days) per local label or per the IP Manual (or SPC). Azacitidine may be administered by SC injection or IV infusion. Alternate dosing schedules to administer the 7 doses to accommodate participant and treatment center availability are allowed.
  The starting dose regimen will be the same as the most recent regimen received on the B1371019 or B1371012 study.
  Glasdegib 50, 75 or 100 mg will be orally administered daily and continuously. The starting dose regimen will be the same as the most recent regimen received on the B1371012 or B1371019 study.
  Interventions: Drug: Glasdegib; Drug: Azacitidine

INTERVENTIONS:
Drug: Glasdegib — 25 mg or 100 mg tablet
  Other Names: PF-04449913
Drug: Azacitidine — 100 mg/vial powder for 25 mg/mL suspension for injection

SUMMARY:
An open-label study available to all eligible participants from Study B1371019 and participants originating from Study B1371012 continuing on study intervention with azacitidine with or without glasdegib.

ELIGIBILITY:
Inclusion Criteria:

* Any participant who continues to demonstrate clinical benefit (as determined by the Principal Investigator) from study treatment with azacitidine with or without glasdegib in this Study or from Study B1371012.
* Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Female participants who are pregnant or breastfeeding (if continuing to receive study intervention);
* Participant has been withdrawn from Study B1371019 and Study B1371012 for any reason (including INT cohort participants required to end study treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- Austria (2):
  - Landeskrankenhaus Salzburg, Universitatsklinik fur Innere Medizin III der PMU, Salzburg
  - Uniklinikum Salzburg, Landeskrankenhaus Salzburg, Salzburg
- Canada (2):
  - Health Sciences Centre, Winnipeg, Manitoba
  - CancerCare Manitoba, Winnipeg, Manitoba
- Czechia (2):
  - Ustavni lekarna, Ostrava - Poruba
  - Klinika hematoonkologie, Ostrava-Poruba
- France (2):
  - CHU de Nantes Hotel Dieu, Nantes
  - CHU de Nantes, Nantes
- Hungary (2):
  - Debreceni Egyetem Klinikai Kozpont Belgyogyaszati Klinika, Hematologia Tanszek, Debrecen
  - Debreceni Egyetem Klinikai Kozpont Belgyogyaszati Klinika, Debrecen
- Italy (2):
  - AOU Ospedali Riuniti Umberto I, G.M. Lancisi, G. Salesi, Clinica Di Ematologia, Torrette Di Ancona, Ancona
  - SOD Farmacia-Dipt dei servizi -AOU Ospedali Riuniti Umberto I, G.M. Lancisi, G. Salesi, Torette Di Ancona, AN
- Japan (2):
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Osaka City University Hospital, Osaka, Osaka
- Instituto Nacional de Cancerología, México, MÉX, Mexico
- WWCOiT im. M. Kopemlka w Lodzl, Lodz, Poland
- Hospital Universitari i Politecnic La Fe, Valencia, Spain
- The Royal Marsden NHS Foundation Trust, Sutton, Surry, United Kingdom

REFERENCES:
- See also: B1371019 (NCT03416179) — https://clinicaltrials.gov/ct2/show/NCT03416179?term=B1371019&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from non-intensive (NINT) cohort of study B1371019 (NCT03416179) or study B1371012 (NCT02367456) were enrolled in this open label, continuation study. A total of 14 participants were enrolled in this study.
Groups:
- Glasdegib + Azacitidine: Participants received glasdegib 100 milligrams (mg) tablet per oral (PO) once a day (QD) in combination with azacitidine 75 mg per meter squared (m^2)/day as subcutaneous (SC) injection or intravenous (IV) infusion for 7 days every 28 days. Treatment continued until objective disease progression or relapse, death, unacceptable toxicity, or participant refusal, whichever occurred first. Participants were followed up for 28 days after end of study treatment.
- Placebo + Azacitidine: Participants received placebo matched to Glasdegib in combination with azacitidine 75mg/m^2/day SC or IV for 7 days every 28 days. Treatment continued until objective disease progression or relapse, death, unacceptable toxicity, or participant refusal, whichever occurred first. Participants were followed up for 28 days after end of study treatment.
Period: Overall Study
Arm/Group | Glasdegib + Azacitidine | Placebo + Azacitidine
Started | 9 | 5
Treated | 8 | 5
Completed | 3 | 1
Not Completed | 6 | 4
Not completed — Death | 1 | 0
Not completed — Other | 4 | 4
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who receive at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Glasdegib + Azacitidine | Placebo + Azacitidine | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.33 (3.94) | 76.80 (5.26) | 73.93 (4.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 7 | 4 | 11
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (AE) and Treatment Related AE
Description: AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. An AE was considered treatment emergent if the event occurred during the on-treatment period (regardless of if it was seen prior to the start of treatment). An AE was considered treatment related as assigned by the investigator.
Time Frame: From initiation of study treatment to study completed from 17-May-2021 to 02-Dec-2022 (approximately 565 days)
Population: Safety analysis set included all participants who receive at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasdegib + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 9 | 5
Participants
  Treatment emergent AE | 7 | 4
  Treatment related AE | 5 | 4

2. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (SAE) and Treatment Related SAEs
Description: A SAE was defined as any untoward medical occurrence that, at any dose that resulted in death; was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect or other medical events as per investigator's judgement. A SAE was considered treatment emergent if the event occurred during the on-treatment period (regardless of if it was seen prior to the start of treatment). A SAE was considered treatment related as assigned by the investigator.
Time Frame: From initiation of study treatment to study completed from 17-May-2021 to 02-Dec-2022 (approximately 565 days)
Population: Safety analysis set included all participants who receive at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Glasdegib + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 9 | 5
Participants
  Treatment emergent SAEs | 2 | 1
  Treatment related SAEs | 1 | 1

ADVERSE EVENTS:
Time Frame: From initiation of study treatment to study completed from 17-May-2021 to 02-Dec-2022 (approximately 565 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Arm/Group | Glasdegib + Azacitidine | Placebo + Azacitidine
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/9 | 1/5
Other Adverse Events (participants affected / at risk) | 6/9 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glasdegib + Azacitidine (N=9) | Placebo + Azacitidine (N=5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Glasdegib + Azacitidine (N=9) | Placebo + Azacitidine (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Corynebacterium bacteraemia (Infections and infestations) | 1 | 0
Epstein-Barr virus infection reactivation (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT04842604/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT04842604/SAP_001.pdf